CLINICAL TRIAL: NCT00193011
Title: A Randomized Multicenter Trial Comparing Weekly Docetaxel and CMF in the Adjuvant Treatment of Women With High-Risk Breast Cancer Who Are > 65 Years Old or Are Not Candidates for Anthracycline-Based Adjuvant Therapy
Brief Title: Weekly Docetaxel and CMF in the Adjuvant Treatment of Elderly Women With High-Risk Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Denise A. Yardley, M.D., Sarah Cannon Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 41; GIA 11169
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Methotrexate; Fluorouracil

ARMS (2):
- 1 (Experimental): Docetaxel
  Interventions: Drug: Docetaxel
- 2 (Experimental): Cyclophosphamide + Methotrexate + 5-fluorouracil
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Docetaxel — Docetaxel
  Arms: 1
Drug: Cyclophosphamide — Cyclophosphamide
  Arms: 2
Drug: Methotrexate — Methotrexate
  Arms: 2
Drug: 5-Fluorouracil — 5-Fluorouracil
  Arms: 2

SUMMARY:
This trial will evaluate the effectiveness of standard adjuvant treatment with CMF chemotherapy versus treatment with weekly docetaxel in patients with high-risk breast cancer who are 65 years of age and older or are poor candidates for anthracycline-containing regimens. This CMF regimen has decreased dose intensity and may be slightly less active in patients with metastatic breast cancer; however, the patient population in this trial has tolerated more intensive CMF regimens poorly in other trials.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

* Docetaxel
* Cyclophosphamide + Methotrexate + 5-fluorouracil

This is not a blinded study so both the patient and the investigator will know which treatment has been assigned.

Chemotherapy will be followed by breast and/or regional radiotherapy in appropriate patients, and by hormone therapy with tamoxifen for 5 years in patients who are estrogen-receptor positive. Patients who are considered poor candidates to receive tamoxifen may receive hormonal therapy with anastrazole.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Female patients with adenocarcinoma of the breast confirmed by biopsy
* Age 65 or older
* Under age 65 must have significant medical illness, or general frailty
* Adequate bone marrow, liver or kidney function
* Normal heart function
* Less than 84 days from mastectomy/lumpectomy or axillary dissection
* Signed consent obtained prior to initiation of any study procedures

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Received neo-adjuvant therapy
* Primary tumor is locally advanced at diagnosis
* Received prior chemotherapy within five years
* Received previous radiation therapy within 5 years
* Peripheral neuropathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-03; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 18 months

SECONDARY OUTCOMES:
overall survival | 18 months
toxicity | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC